CLINICAL TRIAL: NCT03508310
Title: A Waiting Room-Delivered Video to Enhance Antiretroviral Therapy Readiness, Adherence, and Retention in Care for Minority Persons Living With HIV Infection
Brief Title: A Waiting Room-Delivered Video to Enhance Clinical Outcomes Among Persons Living With HIV
Acronym: TCOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Sentient Research (Industry); UCLA David Geffen School of Medicine and Fielding School of Public Health (Unknown); Denver STD Prevention Training Center, Denver Public Health Department (Unknown); California State University, Long Beach (Other); Education Development Center, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1163249
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Quasi-experimental design, in which the intervention condition (i.e., video and posters) was implemented for 10 months and the historical comparison condition (i.e., standard waiting room environment) was the prior 10-month period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 29-minute clinic waiting room video intervention that includes three vignettes and a 2-part animation sequence about main characters who model overcoming challenges to optimal HIV care. The video was played on continuous loop in recognition of typically short patient wait times. Waiting room posters used images from the video to direct patients' attention to the video and reinforce prevention messages.
  Interventions: Other: Taking Care of Me Video
- Comparison (No Intervention): Historical comparison condition. Patients were exposed to standard waiting room environment (absent of intervention video and posters).

INTERVENTIONS:
Other: Taking Care of Me Video — The video's conceptual framework incorporates Social Cognitive Theory, Information-Motivation-Behavioral Skills model, and Social Action Theory, which together address cognitive and behavioral factors related to study outcomes. Storylines embedded prevention messages aimed at increasing treatment initiation (n=9), medication adherence (n=35), retention in care (n=22), partner protection (n=12), and communication with health care providers (n=7).
  Arms: Intervention

SUMMARY:
The purpose of this project is to beta-test a brief waiting room video intervention that promotes early initiation of antiretroviral treatment among treatment-naïve HIV-positive patients, adherence to antiretroviral treatment and retention in care among HIV-positive patients currently on therapy, sexual risk reduction tailored to HIV-positive persons, and patient-initiated discussion of these topics with their health providers. The video is currently being created, and will be ready for beta-testing by June 1, 2016. Results of the beta-testing will be used to refine and improve the video before dissemination to HIV/AIDS treatment facilities nationally. This video project is being funded by the Centers for Disease Control and Prevention, Division of HIV/AIDS Prevention (DHAP).

DETAILED DESCRIPTION:
The overall goal of this study is to beta-test the waiting room video in three HIV/AIDS treatment facilities in different US jurisdictions with high AIDS prevalence. These results will be used to refine the video and to increase its effectiveness among minority persons living with HIV infection. The beta-testing will consist of: 1) unobtrusive observations of waiting room patients for one day at each facility and 2) de-identified, existing patient medical data abstracted from each facility's electronic medical record (EMR) system to investigate outcomes relevant to HIV medication adherence and retention in care.

ELIGIBILITY:
Inclusion Criteria:

HIV/AIDS treatment facility inclusion: The participating treatment facilities will have a combined total of at least 2,700 monthly patient visits during the study period. Each of the HIV/AIDS treatment facilities meets the following inclusion criteria:

1. located in a jurisdiction with high AIDS prevalence;
2. managing more than 500 unique HIV-positive patients annually;
3. serving minority persons such that minimally 55% of the clinic population is African-American and Hispanic/Latino;
4. at least 163 patients have unsuppressed viral load;
5. utilizing an electronic medical record (EMR) system; and
6. not participating in another behavioral intervention research project during the historical comparison data period (August 2015 through May 2016) or during the 10-month intervention period (June 2016 through March 2017).

Exclusion Criteria:

-

Ages: 18 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4003 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Antiretroviral therapy (ART) medication adherence (suppression level) | By 6 months (183 days) after the patient's index (first) visit to the clinic
  Adherence was measured by whether viral load suppression (<200 RNA copies/mL) was achieved
Antiretroviral therapy (ART) medication adherence (undetectable level) | By 6 months (183 days) after the patient's index (first) visit to the clinic
  Adherence was measured by whether viral load suppression (<50 RNA copies/mL) was achieved

SECONDARY OUTCOMES:
Treatment initiation | on, before, or within 7 days after, their index visit, as documented by OAMC visits in patient EMRs.
  Treatment initiation was measured by a patient's receipt of an ART prescription
Retention in HIV medical care | 2 or more clinic visits for any reason at least 90 days apart in the past year divided by all active clients who had had at least one such visit in the past year
  Measured by an adaptation of the Health Resources and Services Administration's (HRSA) definition in the Annual Ryan White HIV/AIDS Program Services Report

CONTACTS AND LOCATIONS:
Overall Officials: Mary S. Neumann, PhD, Principal Investigator — Centers for Disease Control and Prevention; Aaron Plant, MPH, Principal Investigator — Sentient Research

IPD SHARING:
Plan to Share IPD: Yes
When appropriate, data sets will be made available to interested researchers following discussion with study team.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: To be determined
Access Criteria: To be determined

REFERENCES:
- [Derived] Neumann MS, Plant A, Margolis AD, Borkowf CB, Malotte CK, Rietmeijer CA, Flores SA, O'Donnell L, Robilotto S, Myint-U A, Montoya JA, Javanbakht M, Klausner JD. Effects of a brief video intervention on treatment initiation and adherence among patients attending human immunodeficiency virus treatment clinics. PLoS One. 2018 Oct 5;13(10):e0204599. doi: 10.1371/journal.pone.0204599. eCollection 2018. PMID 30289884